CLINICAL TRIAL: NCT01409460
Title: Is an Obturator Nerve Block Required for Every Patient Having Total Knee Arthroplasty With Femoral and Sciatic Nerve Block?
Brief Title: Obturator Nerve Block With Femoral and Sciatic Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sanjay Sinha, Saint Francis Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-10-003
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2008-10

CONDITIONS: Nerve Block; Pain Medication
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- True Obturator Nerve Block (Experimental)
  Interventions: Procedure: Oburator Nerve block
- Sham Block (Sham Comparator)
  Interventions: Procedure: Sham Injection in pectineus muscle.

INTERVENTIONS:
Procedure: Oburator Nerve block — Use of selective pain block.
  Arms: True Obturator Nerve Block
Procedure: Sham Injection in pectineus muscle. — Five minutes after the sham block pain was assessed in these patients. If pain score was 5 or greater a true obturator nerve block was performed on these patients.
  Arms: Sham Block

SUMMARY:
The purpose of this study is to evaluate how many patients require the addition of the obturator nerve block in the recovery room after the total knee surgery. Also to study the efficacy of blocking the obturator nerve in controlling their knee pain.

ELIGIBILITY:
Inclusion Criteria:

* total knee replacement

Exclusion Criteria:

* Hisory of neurologica disease, diabetes, pregnancy, neuropathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To assess the use of obturator Nerve block for patients undergoing total knee arthroplasty | 15 minutes in recovery room post operatively
  The need for rescue obturator nerve block in total knee arthoplasty patients who have sucessful femoral nerve block and sciatic nerve block in place.

SECONDARY OUTCOMES:
Pain medication use intra-operatively and in the recovery room after surgery. Pain scores in recovery room. | During surgery and until discharge from recovery room.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States